CLINICAL TRIAL: NCT00846924
Title: 30-Day Cardiac Event Monitor Belt for Recording Atrial Fibrillation After a Cerebral Ischemic Event: A Randomized Controlled Trial
Brief Title: 30-Day Cardiac Event Monitor Belt for Recording Atrial Fibrillation After a Cerebral Ischemic Event
Acronym: EMBRACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. David Gladstone, Study Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Embrace001
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Stroke; Transient Ischemic Attack; Atrial Fibrillation; Atrial Flutter
Keywords: Stroke; Transient Ischemic Attack; Atrial fibrillation; Atrial flutter
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- repeat 24-hour Holter monitor (Active Comparator)
  Interventions: Device: 24-hour Holter
- 30-day ambulatory cardiac event monitor (Experimental)
  Interventions: Device: a 30-day ambulatory cardiac event monitor

INTERVENTIONS:
Device: a 30-day ambulatory cardiac event monitor — Patients will be fitted with dry electrode belt (including cardiac event monitor)and instructed to wear the device for as many hours(waking and sleeping) each day as possible, for a total of 30 days.
  Other Names: AccuHeart Electrode Belt, Braemar ER 910AF (cardiac event monitor)
  Arms: 30-day ambulatory cardiac event monitor
Device: 24-hour Holter — Repeat standard 24-hour Holter Monitor
  Other Names: Performed as per individual hospital routines
  Arms: repeat 24-hour Holter monitor

SUMMARY:
Atrial fibrillation is the most common cardiac cause of ischemic stroke. Detecting atrial fibrillation after a stroke or TIA is critical because highly effective secondary stroke prevention therapy is available for individuals who are recognized to have atrial fibrillation. However, atrial fibrillation is likely under-diagnosed after stroke and TIA because atrial fibrillation is often difficult to detect as it is frequently paroxysmal and asymptomatic, and patients do not routinely undergo prolonged screening. The purpose of this study is to determine the diagnostic yield of a novel 30-day cardiac event monitor compared to a repeat 24-hour Holter monitor for detecting occult paroxysmal atrial fibrillation in patients with a recent ischemic stroke or TIA of undetermined etiology after completion of a standard clinical stroke work-up (including an initial negative Holter monitor.)

ELIGIBILITY:
Inclusion:

1. Diagnosis of the index event* made by a stroke specialist of an acute ischemic stroke or TIA (WHO definition) of undetermined etiology (cryptogenic) occurring within the previous 6 months (180 days).The event must be either:

   * an embolic arterial ischemic stroke confirmed by neuroimaging; or
   * a transient ischemic attack, defined as involving a focal unilateral motor deficit, speech/language deficit, or hemianopia, with symptom duration <24 hours (note: amaurosis fugax/transient monocular blindness, pure sensory spells, isolated vertigo spells, etc. do not qualify for enrolment given the potential for misdiagnosis of such events).
2. Patient meets the following:

   * At least one 12-lead ECG has already been obtained as part of the routine clinical post-stroke/TIA work-up, and no ECGs have shown any episodes of atrial fibrillation or atrial flutter, and;
   * A Holter monitor has already been obtained as part of the routine clinical post-stroke/TIA work-up, and does not show any episodes of atrial fibrillation or atrial flutter ≥30 seconds.
3. The patient is being actively investigated for the etiology of the stroke/TIA event and additional cardiac monitoring is desired to screen further for the possibility of occult paroxysmal atrial fibrillation/flutter, i.e. patients selected for this study are those for whom the investigator, in his/her clinical judgment, would consider ordering a repeat Holter monitor as part of clinical care.
4. The following diagnostic tests have already been completed as part of clinical routine post-stroke/TIA:

   * brain imaging with CT or MRI,
   * vascular imaging of the extracranial and intracranial circulation with either CT angiography or MR angiography to exclude significant large vessel occlusive disease as the most likely mechanism for the index ischemic event (carotid Doppler ultrasound is acceptable for those presenting with anterior circulation ischemic events),
   * transthoracic (or transesophageal) echocardiography to exclude thrombus or other structural heart disease that in the opinion of the investigator is the most likely cause for the stroke/TIA event. [Note: If a baseline echocardiogram cannot be obtained clinically after the index event and prior to study enrollment, then it is acceptable for study purposes for an echocardiogram to be obtained after patient enrollment into the study but prior to the 90-day follow-up visit. Alternatively, an echocardiogram already performed within one year prior to study enrollment may serve as the baseline echocardiogram for study purposes.]
5. Age 55 years or older [Note: Participants aged 55-59 years should have imaging confirmation of the index stroke/TIA event with an embolic imaging pattern of acute cerebral ischemia]
6. Informed consent from the patient (or from a legally authorized representative if the patient is not competent, e.g. due to stroke-related cognitive impairment, aphasia, or anosognosia).
7. The patient is expected to survive at least 6 months.
8. The patient has a valid provincial health insurance number.

   * The index event will be defined as the event leading to medical presentation

Exclusion:

1. Any previously documented atrial fibrillation or atrial flutter, i.e. a past history of atrial fibrillation/flutter or atrial fibrillation/flutter detected on ECG, Holter, or telemetry following the index stroke/TIA event (a remote history of transient perioperative atrial fibrillation is not exclusionary
2. Exclusively retinal stroke or TIA event.
3. A most responsible etiological diagnosis for the qualifying stroke/TIA event has already been determined, i.e. probable small-vessel (lacunar) disease, probable large vessel disease, cervicocephalic artery dissection, venous sinus thrombosis, hypercoagulable states, or other known cause.
4. Planned carotid endarterectomy within 90 days.
5. Patient is already currently participating in a clinical trial involving an investigational medication or device.*
6. Any finding on echocardiography for which there is already an evidence-based indication for long-term anticoagulation (e.g. mechanical heart valve, thrombus, etc.).
7. Endocarditis
8. Pacemaker or ICD device.
9. Patients with known skin reactions to synthetic polymers or to silver. (Some people who display sensitivity to silver jewellery are sensitive to the impurities present in silver alloys and not to the silver itself. These people may participate.)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2009-05; Primary Completion 2014-04 (Actual); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Detection of one or more episodes of atrial fibrillation or atrial flutter ≥30 seconds, as assessed at the 90 day follow-up | 90 days

SECONDARY OUTCOMES:
Atrial fibrillation <30 seconds | 90 days
Atrial flutter <30 seconds | 90 days
Non-sustained (>3 beats, <30 seconds) irregular atrial tachyarrhythmia (including brief runs of atrial fibrillation) | 90 days
Proportion of patients in each group that are prescribed oral anticoagulation, as assessed at the 90-day follow-up | 90 days
Patient adherence with 30-day monitoring: average proportion of days wearing the monitor per patient, and the percentage of patients wearing the monitor for >75% of the target period | 90 days
1 and 2-year recurrence of ischemic stroke/TIA, death, hemorrhagic stroke, major adverse bleeding event, detection of atrial fibrillation outside of the study protocol | 2 years
composite endpoint of: (1) AF >30 seconds, (2) non-sustained (>3 beats, <30 seconds) irregular atrial tachyarrhythmia (including brief runs of AF), or (3) atrial flutter. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: David J Gladstone, MD, PhD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (17):
- Canada (17):
  - Foothills Medical Centre, Calgary, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Vancouver Hospital and Health Sciences Centre, Vancouver, British Columbia
  - Vancouver Island Health Research Centre (VIHA), Victoria, British Columbia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Robarts Research Institute, London, Ontario
  - Ottawa Hospital Research Institute -The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Regional HSC, Thunder Bay, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - UHN / Toronto Western Hospital, Toronto, Ontario
  - York Central Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - CHA-Hôpital de l'Enfant-Jesus, Québec, Quebec

REFERENCES:
- [Derived] Gladstone DJ, Dorian P, Spring M, Panzov V, Mamdani M, Healey JS, Thorpe KE; EMBRACE Steering Committee and Investigators. Atrial premature beats predict atrial fibrillation in cryptogenic stroke: results from the EMBRACE trial. Stroke. 2015 Apr;46(4):936-41. doi: 10.1161/STROKEAHA.115.008714. Epub 2015 Feb 19. PMID 25700289
- [Derived] Gladstone DJ, Spring M, Dorian P, Panzov V, Thorpe KE, Hall J, Vaid H, O'Donnell M, Laupacis A, Cote R, Sharma M, Blakely JA, Shuaib A, Hachinski V, Coutts SB, Sahlas DJ, Teal P, Yip S, Spence JD, Buck B, Verreault S, Casaubon LK, Penn A, Selchen D, Jin A, Howse D, Mehdiratta M, Boyle K, Aviv R, Kapral MK, Mamdani M; EMBRACE Investigators and Coordinators. Atrial fibrillation in patients with cryptogenic stroke. N Engl J Med. 2014 Jun 26;370(26):2467-77. doi: 10.1056/NEJMoa1311376. PMID 24963566